CLINICAL TRIAL: NCT03693001
Title: Clinical and Morphological Effects of Hyperbaric Oxygen Therapy in Patients With Interstitial Cystitis Associated With Fibromyalgia
Brief Title: HBOT for Patients With IC/FM (Interstitial Cystitis/Fibromyalgia)
Acronym: IC/FMHBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HEC-DSB 07/16 Padua, It
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia; Interstitial Cystitis
MeSH Terms: conditions — Fibromyalgia; Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IC/FM Patients (Experimental): All patients had been diagnosed with fibromyalgia and were suffering from IC by standard criteria.
  Interventions: Device: Intermittent Exposure to Oxygen via Oro-Nasal Mask

INTERVENTIONS:
Device: Intermittent Exposure to Oxygen via Oro-Nasal Mask — Patients were exposed to breathing 100% oxygen at 2 atmospheres absolute (ATA) in a multiplace pressure chamber for 90 minutes using an oro-nasal mask for 40 treatments over a 2 month period.

SUMMARY:
The investigators observed 12 fibromyalgia and interstitial cystitis patients undergoing hyperbaric oxygen oxygen treatment in a multiplace pressure chamber for 90 minutes, 40 treatment each, using an oro-nasal mask.

DETAILED DESCRIPTION:
The investigators structured a prospective observational pilot experimental design in consenting patients with IC and FM, with repeated subjective and urological measures conducted before and after a therapeutic protocol. The study duration was set to 3 months. Patients were exposed to breathing 100% oxygen at 2 atmospheres absolute (ATA) in a multiplace pressure chamber for 90 minutes using an oro-nasal mask. Patients undertook a cycle of 20 sessions for 5 days per week for four weeks. After one week of suspension, a second cycle of 20 sessions was completed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of absence of Hunner's ulcers
* Pain in bladder that improves with urination
* pain(supra-pubic, pelvic, urethral, vaginal, or perineal)
* presence of glomerulation or bleeding +/- at the cystodistension
* reduced capacity
* increased proprioceptive sensitivity
* normal or reduced compliance
* number of tender points that establish that diagnosis

Exclusion Criteria:

* Pregnancy (diagnosed or within a year)
* age less than 18 years
* benign or malignant bladder tumors
* radiation cystitis
* symptomatic bladder diversions
* herpes in active phase
* bladder and urethral stones
* urinary frequency less than 10 times a day
* presence of symptoms less than 12 months
* bladder capacity>400ml with no sensitive urgency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Frequency of Urination | 1-3 months after completing procedure
  Frequency of Urination was measured via a voiding diary. Patients recorded all urinary events via the voiding diary.
Pain symptoms in IC patients | 1-3 months after completing procedure
  Widespread Pain Index (WPI): total amount ranges from 0 to 19 points corresponding to the possibly-painful 19 body areas (i.e., areas of the shoulders, arms, hips, legs, jaws, chest, abdomen, back, and neck).
Pain Symptoms in IC patients | 1-3 months after completing procedure
  Pelvic Pain & Urgency and Frequency Symptom Scale (PUF: Total scores range from 0-35 (symptom subscale 0-23 and bother subscale 0-12). The higher the scores, the more severe the level of symptoms.
Bladder Capacity (as part of symptoms) | 1-3 months after completing procedure
  Symptom Severity Scale (SSS): symptoms are measured on the basis of a 0-3 severity scale considering fatigue, waking unrefreshed, and cognitive symptoms. The greater the amount, the more severe the symptomatology.
Bladder Capacity | 1-3 months after completing procedure
  O'Leary Saint Index: measures the symptoms of the lower urinary tract and their influence on quality-of-life in subjects with IC. Scales range from 0-5 in most cases, with 0 being indicative of little to no symptoms and higher numbers indicative of more severe symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Bosco, MD, Study Director — University of Padova

IPD SHARING:
Plan to Share IPD: Yes
We are planning wide distribution of these results among urologists, neurologists, and internal medicine specialists.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: upon email request.

REFERENCES:
- [Background] Parsons CL, Dell J, Stanford EJ, Bullen M, Kahn BS, Waxell T, Koziol JA. Increased prevalence of interstitial cystitis: previously unrecognized urologic and gynecologic cases identified using a new symptom questionnaire and intravesical potassium sensitivity. Urology. 2002 Oct;60(4):573-8. doi: 10.1016/s0090-4295(02)01829-0. PMID 12385909
- [Background] Tanaka T, Nitta Y, Morimoto K, Nishikawa N, Nishihara C, Tamada S, Kawashima H, Nakatani T. Hyperbaric oxygen therapy for painful bladder syndrome/interstitial cystitis resistant to conventional treatments: long-term results of a case series in Japan. BMC Urol. 2011 May 24;11:11. doi: 10.1186/1471-2490-11-11. PMID 21609485
- [Background] van Ophoven A, Rossbach G, Oberpenning F, Hertle L. Hyperbaric oxygen for the treatment of interstitial cystitis: long-term results of a prospective pilot study. Eur Urol. 2004 Jul;46(1):108-13. doi: 10.1016/j.eururo.2004.03.002. PMID 15183555
- [Background] Lee JD, Lee MH. Increased expression of hypoxia-inducible factor-1alpha and vascular endothelial growth factor associated with glomerulation formation in patients with interstitial cystitis. Urology. 2011 Oct;78(4):971.e11-5. doi: 10.1016/j.urology.2011.05.050. Epub 2011 Aug 2. PMID 21813166
- [Background] Loran OB, Siniakova LA, Seregin AV, Mitrokhin AA, Plesovskii AM, Vinarova NA. [Hyperbaric oxygenation in the treatment of patients with interstitial cystitis: clinical and morphological rationale]. Urologiia. 2011 May-Jun;(3):3-5. Russian. PMID 21874665
- [Background] Mathers MJ, Lazica DA, Roth S. [Non-bacterial cystitis: principles, diagnostics and etiogenic therapy options]. Aktuelle Urol. 2010 Nov;41(6):361-8. doi: 10.1055/s-0030-1262615. Epub 2010 Nov 16. German. PMID 21082515
- [Background] Nickel JC, Tripp DA, Pontari M, Moldwin R, Mayer R, Carr LK, Doggweiler R, Yang CC, Mishra N, Nordling J. Interstitial cystitis/painful bladder syndrome and associated medical conditions with an emphasis on irritable bowel syndrome, fibromyalgia and chronic fatigue syndrome. J Urol. 2010 Oct;184(4):1358-63. doi: 10.1016/j.juro.2010.06.005. Epub 2010 Aug 17. PMID 20719340
- [Background] Efrati S, Golan H, Bechor Y, Faran Y, Daphna-Tekoah S, Sekler G, Fishlev G, Ablin JN, Bergan J, Volkov O, Friedman M, Ben-Jacob E, Buskila D. Hyperbaric oxygen therapy can diminish fibromyalgia syndrome--prospective clinical trial. PLoS One. 2015 May 26;10(5):e0127012. doi: 10.1371/journal.pone.0127012. eCollection 2015. PMID 26010952
- [Background] Arnold LM, Clauw DJ, McCarberg BH; FibroCollaborative. Improving the recognition and diagnosis of fibromyalgia. Mayo Clin Proc. 2011 May;86(5):457-64. doi: 10.4065/mcp.2010.0738. PMID 21531887
- [Background] Yildiz S, Kiralp MZ, Akin A, Keskin I, Ay H, Dursun H, Cimsit M. A new treatment modality for fibromyalgia syndrome: hyperbaric oxygen therapy. J Int Med Res. 2004 May-Jun;32(3):263-7. doi: 10.1177/147323000403200305. PMID 15174219
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Background] Brewer ME, White WM, Klein FA, Klein LM, Waters WB. Validity of Pelvic Pain, Urgency, and Frequency questionnaire in patients with interstitial cystitis/painful bladder syndrome. Urology. 2007 Oct;70(4):646-9. doi: 10.1016/j.urology.2007.06.1089. Epub 2007 Aug 20. PMID 17707887
- [Background] Jones KD, Maxwell C, Mist SD, King V, Denman MA, Gregory WT. Pelvic Floor and Urinary Distress in Women with Fibromyalgia. Pain Manag Nurs. 2015 Dec;16(6):834-40. doi: 10.1016/j.pmn.2015.06.001. Epub 2015 Aug 8. PMID 26259883
- [Background] Lubeck DP, Whitmore K, Sant GR, Alvarez-Horine S, Lai C. Psychometric validation of the O'leary-Sant interstitial cystitis symptom index in a clinical trial of pentosan polysulfate sodium. Urology. 2001 Jun;57(6 Suppl 1):62-6. doi: 10.1016/s0090-4295(01)01126-8. PMID 11378052
- [Background] Ito T, Tomoe H, Ueda T, Yoshimura N, Sant G, Hanno P. Clinical symptoms scale for interstitial cystitis for diagnosis and for following the course of the disease. Int J Urol. 2003 Oct;10 Suppl:S24-6. doi: 10.1046/j.1442-2042.10.s1.7.x. No abstract available. PMID 14641410
- [Background] Tamaki M, Saito R, Ogawa O, Yoshimura N, Ueda T. Possible mechanisms inducing glomerulations in interstitial cystitis: relationship between endoscopic findings and expression of angiogenic growth factors. J Urol. 2004 Sep;172(3):945-8. doi: 10.1097/01.ju.0000135009.55905.cb. PMID 15311005
- [Derived] Bosco G, Ostardo E, Rizzato A, Garetto G, Paganini M, Melloni G, Giron G, Pietrosanti L, Martinelli I, Camporesi E. Clinical and morphological effects of hyperbaric oxygen therapy in patients with interstitial cystitis associated with fibromyalgia. BMC Urol. 2019 Nov 5;19(1):108. doi: 10.1186/s12894-019-0545-6. PMID 31690286